CLINICAL TRIAL: NCT03157219
Title: Manipal Heart Failure Registry (MHFR): A Long Term, Prospective and Descriptive Study of Heart Failure in a Tertiary Care Hospital in South India
Brief Title: Manipal Heart Failure Registry (MHFR)
Acronym: MHFR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manipal University (Other)
Responsible Party: Principal Investigator, Ajit Singh, PhD, Principal Investigator, Manipal University
Other Study IDs: MUEC/20/2015-16
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure; Systolic Heart Failure; Diastolic Heart Failure; Decompensated Heart Failure; Acute Heart Failure
Keywords: Heart failure; Institutional level registry; Systolic heart failure; Acute heart failure; Heart failure India
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Burden of HF in India is approximate 2-5 million patients with an estimated prevalence of 2-3/1000 population. HF is responsible for approx1.8 million admissions annually in India. Very few studies are there in India which shows the detailed documentation of HF.

Manipal Heart failure Registry (MHFR) is an institutional level Heart Failure disease registry. In MHFR the investigator will document the detailed information about heart failure patients admitted or referred to Department of Cardiology, Kasturba Medical College, a constituent college and teaching hospital of Manipal University.

MHFR will include cohorts of patients with acute heart failure (AHF), with the intention of implementing a long-term follow-up, the use of health economic assessment to evaluate the degree of resource utilization; and quantifying the burden on quality of life for patients. Utilization of drug in HF patients will be evaluated as a part of this study to prevent the use of inappropriate drug therapy and to improve overall drug effectiveness and outcomes. Hence the protocol sought to identify the characteristics and long-term outcomes of Indian patients with acute heart failure admitted in an Indian tertiary care center in South India.

There are no risks to patients participating in the registry study, as standard of care quality will not be affected. It is unlikely that there will be any direct benefit as a result of participation in the HF-disease registry. However, the information contained within this non-interventional registry study will be used for research studies directed at improving the knowledge and treatment of acute heart failure as well as improving patients treatment in the future.

The potential impact of proposed research (Manipal Heart Failure Registry) is envisioned to be four-fold:

1. to enable a broad overview of the routine medical practices for HF treatment;
2. to assess the healthcare resource utilization and drug utilization review for heart failure patients
3. to assess the burden of disease (mortality, re-hospitalization) in the long term; and
4. to provide a novel overview of the impact of HF syndrome on quality of life as well as health economics.

DETAILED DESCRIPTION:
RESEARCH GAPS IDENTIFIED:

Only a couple of registry studies in India have followed patients for not more than one year and therefore long-term data on disease management and healthcare resource utilization and health economics has never addressed adequately. Typically, these studies have focused primarily upon inpatient HF clinical profiles, where detailed long-term documentation of cardiac function, treatment patterns, and outcomes is lacking.

HYPOTHESES:

Long term follow up of heart failure patients can identify the disease characteristics, clinical outcomes and help in the development of a disease progression model, thereby eventually improving the practice standards. Proper utilization of healthcare resources decrease in-hospital and follow up mortality in heart failure patients.

The study team also hypothesize that the commonest cause of acute heart failure in our population in present era is myocardial infarction.

MATERIALS AND METHODS:

This proposed observational study is a single center HF-disease registry that will document the routine patterns of diagnosis and medical care for heart failure as well as treatment type, long-term HF-related clinical events, and re-admission rates following the acute admission index event. In addition to the long-term data collection, the study will also link treatment plans and clinical outcomes, to identify best practice in the HF treatment, as well as extent of healthcare resources use. The registry will also collect data on health-related quality of life.

Eligible patients and caregivers may only be included in the study after providing written (witnessed, where required by law or regulation), IRB/IEC-approved informed consent, or, if incapable of doing so, after such consent has been provided by a legally acceptable representative of the patient.

RISKS AND BENEFITS There are no risks to patients participating in the registry study, as standard of care quality will not be affected. It is unlikely that there will be any direct benefit as a result of participation in the HF-disease registry. However, the information contained within this non-interventional registry study will be used for research studies directed at improving the knowledge and treatment of acute heart failure as well as improving patients' treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 year old, and above
2. Patients with a documented diagnosis of Acute heart failure (or chronic heart failure with acute exacerbations) as decided by the physician according to local practices and their clinical judgment (i.e., History/examination; Chest X-ray; ECG, Echocardiogram, BNP or NT-proBNP).

Exclusion Criteria:

1. Patient's participation in any other clinical trial with an investigational treatment.
2. Use of investigational drugs within 5 half-lives of enrolment, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer (as guideline, last dose for small molecules should have occurred more than 30 days, and for biologics more than 4 months prior to enrolment).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The registry will include adult patients (age >18 years) diagnosed with acute-HF with or without co-morbidities at the time of hospitalization
  No specific population required
  Asian race
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2018-09-09 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Prognosis of Heart Failure | "through study completion, an average of 1 year"
  Post discharge events are measured using symptoms and treatment outcomes assessment at follow up
Characterization of Heart failure | "through study completion, an average of 1 year"
  Characterization of HF is measured using in-hospital assessment at index hospitalization and discharge

SECONDARY OUTCOMES:
Treatment Pattern | "through study completion, an average of 1 year"
  Treatment policies for acute heart failure at admission, during hospital stay and at follow ups
Health care resources utilization | "through study completion, an average of 1 year"
  disease burden and economic burden of disease

OTHER OUTCOMES:
Health related quality of life | "through study completion, an average of 1 year"
  Using patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tom Devasia, MD, DM, FACC, Study Chair — Manipal University; Ajit Singh, PHARM D, PhD, Principal Investigator — Manipal University
Locations (1):
- Dr. Ajit Singh, Manipal, Karnataka, India

IPD SHARING:
Plan to Share IPD: No